CLINICAL TRIAL: NCT04429100
Title: Assessment of Fibrosis by Non-invasive Quantitative Imaging of Collagen in the Liver Using Breath-hold MRI With Comparison With MR Elastography and Liver Biopsy
Brief Title: Rapid Breath-hold Quantitative Macromolecular Proton Fraction Imaging for Liver Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chen Weitian, Professor, Chinese University of Hong Kong
Other Study IDs: 2019.660
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Liver Fibrosis
Keywords: magnetic resonance imaging; quantitative imaging; spin-lock
MeSH Terms: conditions — Liver Cirrhosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- liver fibrosis stage F0
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- early-stage liver fibrosis (F1-2)
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- late-stage liver fibrosis (F3-4)
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — One novel MRI sequence, i.e. the quantitative imaging of macromolecular proton fraction (MPF), will be introduced into this study. MPF is defined as the relative amount of protons associated with macromolecules involved in magnetization exchange with free water protons. This parameter is independent of the pool model used for quantification and the pulse sequences used for data acquisition. Recent studies have found a strong association between MPF and collagen content in the fibrotic liver, indicating MPF is a potential biomarker of early-stage liver fibrosis.

SUMMARY:
Chronic liver disease is a major health problem worldwide. Liver fibrosis is a key feature in most chronic liver diseases. When identified early, liver fibrosis may be reversible. Currently, liver biopsy is the gold standard for the diagnosis of liver fibrosis. Liver biopsy; however, is invasive. Non-invasive diagnostic tools are increasingly used in clinical practice. However, the existing noninvasive methods still have significant limitations to detect early-stage liver fibrosis.

Liver fibrosis is characterized by excessive deposition of collagen-rich connective tissues in the liver. The macromolecular proton fraction (MPF) is an MRI parameter which characterizes the magnetization transfer (MT) effect in tissues. Quantitative MPF imaging is non-invasive and can be used to measure collagen deposition in the liver due to the strong MT effect of collagen. It has been reported MPF quantification can be used for diagnosis of early-stage liver fibrosis. However, the existing approaches require B1, B0, and T1 map in addition to the imaging data for MPF quantification, which makes it challenging to adopt them for routine clinical use.

The investigators propose a fast and robust MPF quantification approach. In contrast to the existing methods which rely on saturation radiofrequency pulses for MPF quantification, our approach is based on spin-lock radiofrequency pulses which have minimum Rabi oscillations. The whole imaging data can be acquired within a breath-hold less than 8 seconds. Our approach only needs a B1 map in addition to the imaging data for MPF quantification. The preliminary clinical studies on 3.0T MRI show the measurement using our approach is specific to collagen content and can be used to detect early-stage liver fibrosis. To further confirm the clinical value of the proposed approach, the investigators will investigate the relationship of the collagen content measured using the proposed non-invasive imaging approach and those measured based on morphometry analysis of histology, and determine the diagnostic value of the proposed method for detection of early stage liver fibrosis in a large cohort. The investigators will also perform comparative studies of the proposed method and the state-of-the-art quantitative MPF imaging technique.

This project will provide a diagnostic technology for early detection of liver fibrosis. The proposed MRI technology also has potential to be used for other clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient group

   * patients with histology-proven liver fibrosis, including those with liver fibrosis stage F0, early-stage liver fibrosis (F1-2), and late stage.

   liver fibrosis(F3-4).
   * patient aged 18 years old and above.
2. Healthy control group

   * controls aged 18 years old and above.

Exclusion Criteria:

* Contraindications to MRI, such as cardiac pacemaker, claustrophobia, pregnancy, metallic implants not suitable for MRI scan.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patients referred to hepatology center affiliated to The Chinese University of Hong Kong (CUHK) will be enrolled in this study. The research team led by one hepatologist as one of our collaborators will be responsible for patient recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 3 years
  diagnostic accuracy of quantitative macromolecular proton fraction imaging based on spin-lock (MPF-SL) for detecting early-stage liver fibrosis.

SECONDARY OUTCOMES:
correlation coefficient | 3 years
  correlations between the MPF quantification and the morphometric scores

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandrin L, Fourquet B, Hasquenoph JM, Yon S, Fournier C, Mal F, Christidis C, Ziol M, Poulet B, Kazemi F, Beaugrand M, Palau R. Transient elastography: a new noninvasive method for assessment of hepatic fibrosis. Ultrasound Med Biol. 2003 Dec;29(12):1705-13. doi: 10.1016/j.ultrasmedbio.2003.07.001. PMID 14698338
- [Background] Yin M, Talwalkar JA, Glaser KJ, Manduca A, Grimm RC, Rossman PJ, Fidler JL, Ehman RL. Assessment of hepatic fibrosis with magnetic resonance elastography. Clin Gastroenterol Hepatol. 2007 Oct;5(10):1207-1213.e2. doi: 10.1016/j.cgh.2007.06.012. PMID 17916548
- [Background] Huwart L, Sempoux C, Vicaut E, Salameh N, Annet L, Danse E, Peeters F, ter Beek LC, Rahier J, Sinkus R, Horsmans Y, Van Beers BE. Magnetic resonance elastography for the noninvasive staging of liver fibrosis. Gastroenterology. 2008 Jul;135(1):32-40. doi: 10.1053/j.gastro.2008.03.076. Epub 2008 Apr 4. PMID 18471441
- [Background] Heye T, Yang SR, Bock M, Brost S, Weigand K, Longerich T, Kauczor HU, Hosch W. MR relaxometry of the liver: significant elevation of T1 relaxation time in patients with liver cirrhosis. Eur Radiol. 2012 Jun;22(6):1224-32. doi: 10.1007/s00330-012-2378-5. Epub 2012 Feb 3. PMID 22302503
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Faria SC, Ganesan K, Mwangi I, Shiehmorteza M, Viamonte B, Mazhar S, Peterson M, Kono Y, Santillan C, Casola G, Sirlin CB. MR imaging of liver fibrosis: current state of the art. Radiographics. 2009 Oct;29(6):1615-35. doi: 10.1148/rg.296095512. PMID 19959511
- [Background] Tan CH, Venkatesh SK. Magnetic Resonance Elastography and Other Magnetic Resonance Imaging Techniques in Chronic Liver Disease: Current Status and Future Directions. Gut Liver. 2016 Sep 15;10(5):672-86. doi: 10.5009/gnl15492. PMID 27563019
- [Background] Imajo K, Kessoku T, Honda Y, Tomeno W, Ogawa Y, Mawatari H, Fujita K, Yoneda M, Taguri M, Hyogo H, Sumida Y, Ono M, Eguchi Y, Inoue T, Yamanaka T, Wada K, Saito S, Nakajima A. Magnetic Resonance Imaging More Accurately Classifies Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease Than Transient Elastography. Gastroenterology. 2016 Mar;150(3):626-637.e7. doi: 10.1053/j.gastro.2015.11.048. Epub 2015 Dec 8. PMID 26677985
- [Background] Park CC, Nguyen P, Hernandez C, Bettencourt R, Ramirez K, Fortney L, Hooker J, Sy E, Savides MT, Alquiraish MH, Valasek MA, Rizo E, Richards L, Brenner D, Sirlin CB, Loomba R. Magnetic Resonance Elastography vs Transient Elastography in Detection of Fibrosis and Noninvasive Measurement of Steatosis in Patients With Biopsy-Proven Nonalcoholic Fatty Liver Disease. Gastroenterology. 2017 Feb;152(3):598-607.e2. doi: 10.1053/j.gastro.2016.10.026. Epub 2016 Oct 27. PMID 27911262
- [Background] Castera L, Foucher J, Bernard PH, Carvalho F, Allaix D, Merrouche W, Couzigou P, de Ledinghen V. Pitfalls of liver stiffness measurement: a 5-year prospective study of 13,369 examinations. Hepatology. 2010 Mar;51(3):828-35. doi: 10.1002/hep.23425. PMID 20063276
- [Background] Arena U, Vizzutti F, Corti G, Ambu S, Stasi C, Bresci S, Moscarella S, Boddi V, Petrarca A, Laffi G, Marra F, Pinzani M. Acute viral hepatitis increases liver stiffness values measured by transient elastography. Hepatology. 2008 Feb;47(2):380-4. doi: 10.1002/hep.22007. PMID 18095306
- [Background] Stikov N, Keenan KE, Pauly JM, Smith RL, Dougherty RF, Gold GE. Cross-relaxation imaging of human articular cartilage. Magn Reson Med. 2011 Sep;66(3):725-34. doi: 10.1002/mrm.22865. Epub 2011 Mar 17. PMID 21416504
- [Background] Sritanyaratana N, Samsonov A, Mossahebi P, Wilson JJ, Block WF, Kijowski R. Cross-relaxation imaging of human patellar cartilage in vivo at 3.0T. Osteoarthritis Cartilage. 2014 Oct;22(10):1568-76. doi: 10.1016/j.joca.2014.06.004. PMID 25278066
- [Background] Yarnykh VL, Tartaglione EV, Ioannou GN. Fast macromolecular proton fraction mapping of the human liver in vivo for quantitative assessment of hepatic fibrosis. NMR Biomed. 2015 Dec;28(12):1716-25. doi: 10.1002/nbm.3437. Epub 2015 Oct 27. PMID 26503401
- [Background] Sled JG, Pike GB. Quantitative imaging of magnetization transfer exchange and relaxation properties in vivo using MRI. Magn Reson Med. 2001 Nov;46(5):923-31. doi: 10.1002/mrm.1278. PMID 11675644
- [Background] Ramani A, Dalton C, Miller DH, Tofts PS, Barker GJ. Precise estimate of fundamental in-vivo MT parameters in human brain in clinically feasible times. Magn Reson Imaging. 2002 Dec;20(10):721-31. doi: 10.1016/s0730-725x(02)00598-2. PMID 12591568
- [Background] Yarnykh VL. Pulsed Z-spectroscopic imaging of cross-relaxation parameters in tissues for human MRI: theory and clinical applications. Magn Reson Med. 2002 May;47(5):929-39. doi: 10.1002/mrm.10120. PMID 11979572
- [Background] Gochberg DF, Gore JC. Quantitative magnetization transfer imaging via selective inversion recovery with short repetition times. Magn Reson Med. 2007 Feb;57(2):437-41. doi: 10.1002/mrm.21143. PMID 17260381
- [Background] Gloor M, Scheffler K, Bieri O. Quantitative magnetization transfer imaging using balanced SSFP. Magn Reson Med. 2008 Sep;60(3):691-700. doi: 10.1002/mrm.21705. PMID 18727085
- [Background] Helms G, Hagberg GE. In vivo quantification of the bound pool T1 in human white matter using the binary spin-bath model of progressive magnetization transfer saturation. Phys Med Biol. 2009 Dec 7;54(23):N529-40. doi: 10.1088/0031-9155/54/23/N01. Epub 2009 Nov 11. PMID 19904029
- [Background] Soellinger M, Langkammer C, Seifert-Held T, Fazekas F, Ropele S. Fast bound pool fraction mapping using stimulated echoes. Magn Reson Med. 2011 Sep;66(3):717-24. doi: 10.1002/mrm.22846. Epub 2011 Mar 24. PMID 21437973
- [Background] Yarnykh VL. Fast macromolecular proton fraction mapping from a single off-resonance magnetization transfer measurement. Magn Reson Med. 2012 Jul;68(1):166-78. doi: 10.1002/mrm.23224. Epub 2011 Dec 21. PMID 22190042
- [Background] Nehrke K, Bornert P. DREAM--a novel approach for robust, ultrafast, multislice B(1) mapping. Magn Reson Med. 2012 Nov;68(5):1517-26. doi: 10.1002/mrm.24158. Epub 2012 Jan 17. PMID 22252850
- [Background] Wong GL, Wong VW, Choi PC, Chan AW, Chum RH, Chan HK, Lau KK, Chim AM, Yiu KK, Chan FK, Sung JJ, Chan HL. Assessment of fibrosis by transient elastography compared with liver biopsy and morphometry in chronic liver diseases. Clin Gastroenterol Hepatol. 2008 Sep;6(9):1027-35. doi: 10.1016/j.cgh.2008.02.038. Epub 2008 May 5. PMID 18456573